CLINICAL TRIAL: NCT05285943
Title: A Comparative Study Between Topical Betamethasone Cream or Topical Olive Oil Cream in Prophylaxis Against Acute Radiodermatitis in Breast Cancer Patients.
Brief Title: Use of Topical Olive Oil Cream for Prophylaxis Against Acute Radiodermatitis in Breast Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Farghali Farid, Professor, Head of Clinical Pharmacy Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CL 2775
Record Dates: First submitted 2021-06-21; First posted 2022-03-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Radiodermatitis; Acute
Keywords: Acute Radiodermatitis; Breast Cancer; Olive Oil
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Betamethasone cream (Active Comparator): Patients will apply Betamethasone Valerate 0.1% cream to the irradiated area twice a day.
  Interventions: Drug: Betamethasone Valerate Cream
- Olive oil cream (Active Comparator): Patients will apply prepared Olive Oil cream to the irradiated area twice a day.
  Interventions: Drug: Olive oil cream
- Base cream (Placebo Comparator): Patients will apply prepared base cream to the irradiated area twice a day.
  Interventions: Other: Base Cream

INTERVENTIONS:
Drug: Olive oil cream — Olive oil prepared in a base cream to be applied to irradiated areas.
  Arms: Olive oil cream
Drug: Betamethasone Valerate Cream — Betamethasone valerate prepared in a base cream to be applied to irradiated areas.
  Arms: Betamethasone cream
Other: Base Cream — The base cream used for preparation of both the betamethasone valerate cream and olive cream will be used as a placebo control to be applied to irradiated areas.
  Arms: Base cream

SUMMARY:
This study aims to compare the prophylactic effect of topical betamethasone valerate cream and topical olive oil cream in the prevention of acute radiation dermatitis (ARD) in breast cancer patients treated with radiation. Betamethasone valerate, olive oil cream and the base cream will be compared in a randomized trial to evaluate and compare the development and degree of ARD grading according to Radiation Toxicity Grading (RTOG) skin toxicity score, percentage of patients with the maximum observed ARD grade for each arm of the study, percentage of patients with moist desquamation for each arm of the study, percentage of radiodermatitis-free patients at end of therapy (EOT=time point specifically at end of 2 weeks post radiation therapy). In addition, the patients' quality of life will be evaluated using Dermatology Life Quality Index (DLQI).

DETAILED DESCRIPTION:
Aim of the study:

* This study will be conducted to compare the efficacy of topical steroid cream and topical olive oil cream instituted from the start of radiotherapy in the prevention of acute radiation dermatitis in breast cancer patients.

Objectives:

1. To compare the prophylactic effect of topical betamethasone valerate cream and topical olive oil cream in the prevention of acute radiation dermatitis in breast cancer patients.
2. To provide prospective data evaluating the quality of life (QoL), as most data on QoL in breast cancer patients are derived from cross-sectional studies.

   Methodology:

   Study Design:

   • This is a prospective, double blinded, randomized, parallel study.

   Study subjects:

   A total of 132 (120 + 12) participants will be recruited in order to achieve a statistical power of 0.8, using an alpha of 0.05.Sample size calculation was performed a priori using G-Power v 3.1. based on multiple comparisons of proportions using Chi-square (χ2) test. The maximal intensity of dermatitis during treatment will be measured in each group in the three groups. The calculations will be based on the effect size of 0.284, defined by Cramer's V as medium effect .

   • The recruited patients will be randomly distributed into three groups: Group 1: Patients will apply betamethasone valerate 0.1% cream to the irradiated area twice a day.

   Group 2: Patients will apply prepared olive oil cream to the irradiated area twice a day.

   Group 3 : Patients will apply prepared base cream to the irradiated area twice a day.
   * The three different creams will have the same base .
   * All applications of the creams will be started at the initiation of radiation therapy. Creams will be applied seven days a week during the radiation therapy period, and continued for two weeks after the completion of radiation therapy. The application of the cream will be after the radiation session and 12 hours later, and in the radiation free days the patient will apply every 12 hours.
   * If the patient develops ARD she will continue our prophylactic creams while taking her medical treatment according to the grade of ARD.
   * Those patients that meet the inclusion criteria will be invited to participate before beginning their radiotherapy process (T0) and data will be collected. Data related to treatment will be obtained from the patients' medical records.

   The data to be collected:
   * Age,
   * marital status,
   * schooling,
   * smoker or non-smoker,
   * Fitzpatrick skin type, which reflects skin complexion and sensitivity to sun Type l; always sunburn/never sun tan, Type 2; always sunburn/little sun tan, Type 3; sometimes sunburn/always sun tan, Type 4; never sunburn/always sun tan ,
   * breast size (full bust circumference),
   * body mass index (BMI),
   * comorbidities,
   * the pathological stage,
   * left or right breast cancer,
   * surgery,
   * previous chemotherapy and type of regimen,
   * Radiotherapy-related variables (Radiotherapy field distribution, number of fields of radiation, total prescribed dose, daily dose, energy of radiation).

     * Patients will be evaluated weekly during the radiation therapy (3-6 weeks) and 2 weeks after the radiation therapy at the following times :

   T1 = 7 days after beginning treatment +/- 3 days; T2 = 14 days after beginning treatment +/- 3 days; T3 = 21 days after beginning treatment +/- 3 days; T4 = 28 days after beginning treatment+/- 3 days; T5 = 35 days after beginning treatment+/- 3 days; T6 = 42 days after beginning treatment+/- 3 days; T7 = 49 days after beginning treatment+/- 3 days. T8 = 56 days after beginning treatment+/- 3 days.

   • The Radiation Therapy Oncology Group (RTOG) scale will be used to classify skin toxicity , Grade 0: being no change; Grade 1: follicular, faint, or dull erythema/epilation/dry desquamation/ decreased sweating; Grade 2: tender or bright erythema, patchy moist desquamation/moderate edema; Grade 3: confluent, moist desquamation other than skin folds, pitting edema; Grade 4: ulceration, hemorrhage, necrosis.

   • To evaluate the impact caused by radiodermatitis, we will use a validated Arabic questionnaire Dermatology Life Quality Index (DLQI).

   Patient Consent:

   • An informed written consent will be taken from all patients. The form will be explained to each patient or her caregiver before asking them to sign it.

   Outcomes to be evaluated:
   * Development and degree of ARD grading according to Radiation Toxicity Grading (RTOG) skin toxicity score {T1=7 days after beginning treatment +/- 3 days; to T8=56 days after beginning treatment+/- 3 days}.

     -Percentage of patients with the maximum observed ARD grade for each arm of the study ,

     -Percentage of patients with moist desquamation for each arm of the study [20],

     -Frequencies of different ARD grades at each time point [18],

     -Percentage of patients radiodermatitis free at end of therapy (EOT=time point specifically at end of 2 weeks post radiation therapy),

     - Mean ARD grade at the different observation time points for each group .

     -Time of development of acute radiodermatitis .
   * Patients quality of life will be measured using an Arabic version of validated questionnaire {T1=7 days after beginning treatment +/- 3 days to T8=56 days after beginning treatment+/- 3 days} .
   * Patients 'subjective symptoms (itching, pain, and burning) will be reported weekly during radiation therapy by patients using a visual analog scale (VAS) (10 cm in length, 0 = no symptoms, 10 = worst possible symptoms). In the analysis VAS recordings will be calculated as sum scores and will be grouped as follows: 0 (no); 1-10 (mild), 11-20 (moderate) and 21-30 (severe symptoms) .
   * Patients evaluation of the treatment satisfaction will be measured by the Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General (FACIT-TS-G) at end of therapy (EOT=time point specifically at end of 2 weeks post radiation therapy) .
   * Percentage of patients with secondary skin infection / need of topical and systemic antibiotics during the whole study.
   * Patients' preference to the creams regarding smell, stickiness and easiness to rub out will be recorded using a visual analog scale (VAS) at end of therapy (EOT=time point specifically at end of 2 weeks post radiation therapy).

   Statistical analysis
   * Statistics of the study population will be described using sums and proportions. Chi-square (χ2) test will be used to calculate effect of treatment on skin reaction for categorical data.
   * A two-tailed P value < 0.05 will be deemed statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast malignancy,
* Surgical intervention for carcinoma of the breast with or without lymph node metastasis.
* Treatment with planned course of radiation therapy 5 days a week for 3-6 weeks.
* Good Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1).
* Total radiation dose of ≥42 Gy.

Exclusion Criteria:

* Pregnant and lactating mothers.
* Previous radiation to the chest or breast area.
* Concomitant chemotherapy.
* Concomitant medication that may cause skin reactions.
* Use of any other product on the skin at the treatment site at any time of the study.
* Active dermatitis, history of autoimmune and connective tissue diseases, skin inflammatory diseases or any other specific skin disease.
* Treatment with local or oral corticosteroid, or antioxidant medications.
* Allergy to olive oil.
* Inflammatory carcinoma of the breast as well as those with a known allergy to olive oil.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Acute Radiation Dermatitis (ARD) grading | T1=7 days after beginning treatment +/- 3 days; to T8=56 days after beginning treatment+/- 3 days}.
  • Development and degree of ARD grading according to Radiation Toxicity Grading (RTOG) skin toxicity score

SECONDARY OUTCOMES:
Quality of Life questionnaire | {T1=7 days after beginning treatment +/- 3 days to T8=56 days after beginning treatment+/- 3 days} .
  Patients quality of life will be measured using an Arabic version of a validated questionnaire
Patient Satisfaction | Two weeks post the last dose of radiation therapy
  Patients evaluation of the treatment satisfaction will be measured by the FACIT-TS-G

OTHER OUTCOMES:
Subjective Symptoms | Weekly During Radiation Therapy up to 8 weeks
  Patients 'subjective symptoms (itching, pain, and burning) will be reported using a visual analog scale (VAS) (10 cm in length, 0 = no symptoms, 10 = worst possible symptoms). In the analysis VAS recordings will be calculated as sum scores and will be grouped as follows: 0 (no); 1-10 (mild), 11-20 (moderate) and 21-30 (severe symptoms) .
Skin Infections During Treatment | During the whole study (from recruitment and as long as patient is receiving radiation therapy)up to 8 weeks
  • Percentage of patients with secondary skin infection / need of topical and systemic antibiotics

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McQuestion M. Evidence-based skin care management in radiation therapy: clinical update. Semin Oncol Nurs. 2011 May;27(2):e1-17. doi: 10.1016/j.soncn.2011.02.009. PMID 21514477
- [Background] Fuzissaki MA, Paiva CE, Oliveira MA, Lajolo Canto PP, Paiva Maia YC. The Impact of Radiodermatitis on Breast Cancer Patients' Quality of Life During Radiotherapy: A Prospective Cohort Study. J Pain Symptom Manage. 2019 Jul;58(1):92-99.e1. doi: 10.1016/j.jpainsymman.2019.03.017. Epub 2019 Apr 8. PMID 30974233
- [Background] Ulff E, Maroti M, Serup J, Falkmer U. A potent steroid cream is superior to emollients in reducing acute radiation dermatitis in breast cancer patients treated with adjuvant radiotherapy. A randomised study of betamethasone versus two moisturizing creams. Radiother Oncol. 2013 Aug;108(2):287-92. doi: 10.1016/j.radonc.2013.05.033. Epub 2013 Jul 2. PMID 23827771
- [Background] Cui Z, Xin M, Yin H, Zhang J, Han F. Topical use of olive oil preparation to prevent radiodermatitis: results of a prospective study in nasopharyngeal carcinoma patients. Int J Clin Exp Med. 2015 Jul 15;8(7):11000-6. eCollection 2015. PMID 26379896
- [Background] Ulff E, Maroti M, Serup J, Nilsson M, Falkmer U. Prophylactic treatment with a potent corticosteroid cream ameliorates radiodermatitis, independent of radiation schedule: A randomized double blinded study. Radiother Oncol. 2017 Jan;122(1):50-53. doi: 10.1016/j.radonc.2016.11.013. Epub 2016 Nov 29. PMID 27913066
- [Background] Peipert JD, Beaumont JL, Bode R, Cella D, Garcia SF, Hahn EA. Development and validation of the functional assessment of chronic illness therapy treatment satisfaction (FACIT TS) measures. Qual Life Res. 2014 Apr;23(3):815-24. doi: 10.1007/s11136-013-0520-8. Epub 2013 Sep 24. PMID 24062239
- [Derived] Mohamed IK, Abbassi MM, Kelany MR, Farid SF. Efficacy of Topical Betamethasone Valerate and Olive Oil in Preventing Acute Radiation Dermatitis in Breast Cancer: A Randomized Double-Blind Placebo-Controlled Study. Clin Breast Cancer. 2026 Jan;26(1):348-359.e1. doi: 10.1016/j.clbc.2025.08.008. Epub 2025 Aug 21. PMID 40973558